CLINICAL TRIAL: NCT01193647
Title: Genetic Factors Affecting Risks for Rotator Cuff Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Robert Tashjian, M.D., University of Utah
Other Study IDs: 29048
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Studying the Genetic Relationship of Rotator Cuff Tears

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA will be retained
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will begin to evaluate the heritability of rotator cuff disease, and begin creation of a powerful resource for future genetic studies of rotator cuff disease.

DETAILED DESCRIPTION:
Aim 1. We will recruit and study all patients of the PI who undergo MRI for shoulder complaints. The PI is a shoulder and elbow surgeon and treats a variety of shoulder and non-shoulder pathology. All patients agreeing to participate will undergo a history, physical examination of the shoulder, recording of demographics, family history, genealogy, and risk factors. All participants will provide a blood or saliva sample. Serum and DNA will be stored at the University of Utah for future analysis. Based upon the results of MRI, patients will be categorized based on the presence or absence or rotator cuff tearing. We hope to extend to hospital-wide ascertainment eventually. All patients will be asked if they have known cases of shoulder disorders in their family members. Patients will have the option of sharing their living family members name and contact information with the research team, so we can contact them and invite them to the study.

Aim 2. From this DNA bio-repository, we will begin to describe the familial nature of rotator cuff disease and the characteristics related to increased risk. We will also begin ascertainment and sampling of high-risk individuals and pedigrees, perform association studies to identify risk-associated variants, and screen candidate genes as funding is available.

Aim 3: Utilizing the Utah Population Database (UPDB), we will also define high risk pedigrees within the cohort of individuals with rotator cuff tears. We will also use the database to identify high risk pedigrees by examining the information on family members of patients of with tears to identify high risk pedigrees as well. The RGE has already approved the use of the UPDB for these purposes.

Aim 4: Use UUHSC medical records linked to the UPDB to define the heritable nature of rotator cuff injury and other tendonopathies.

Aim 5: Determine ABO frequencies for patients with rotator cuff tears and compare to population normals utilizing the UPDB.

Aim 6: Use UUHSC medical records linked to the UPDB to define the heritable nature of rotator cuff injury and compression neuropathies.

Aim 7: Query the UUHSC EDW for rotator cuff repair codes and obtain the ABO blood typing for these patients. We will also obtain operative room reports, names and MRN numbers for these patients to ensure there aren't duplications between already enrolled patients and UUHSC EDW findings.

ELIGIBILITY:
Inclusion Criteria:

* Includes any patient who has had a shoulder MRI performed to evaluate shoulder pain as part of a standard clinical exam.
* All first degree relatives of patients with documented rotator cuff tearing will also be possible study participants.
* All patients of Drs. Tashjian, Burks and Greis who have undergone surgical rotator cuff repair.

Exclusion Criteria:

* Exclude any patient who has undergone prior shoulder surgery besides surgery performed by the PI where accurate information, including MRI data exist, regarding the presence or absence of rotator cuff tearing before the surgery.
* Any patient who is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The initial set of study participants for this study will be recruited through the clinical practice of the PI. Patients will be categorized based upon MRI confirmation of a rotator cuff tear. All patients being treated for shoulder pain with a positive MRI for a rotator cuff tear which was performed as a normal part of a clinical exam will be included as possible participants (tear group). All patients being treated for shoulder pain with a negative MRI for rotator cuff tearing (MRI performed for normal part of clinical exam) will undergo an MRI of the opposite shoulder to confirm the absence (or presence) of rotator cuff pathology and be categorized based upon the findings (either tear or no tear group).
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-07; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
evaluate the heritability of rotator cuff disease | 6 years
  All patients agreeing to participate will undergo a history, physical examination of the shoulder, recording of demographics, family history, genealogy, and risk factors. All participants will provide a blood or saliva sample. Serum and DNA will be stored at the University of Utah for future analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Z Tashjian, MD, Principal Investigator — University of Utah Orthopaedic Center
Locations (2):
- United States (2):
  - University of Utah Orthopaedic Center, Salt Lake City, Utah
  - VA Salt Lake City, Salt Lake City, Utah